CLINICAL TRIAL: NCT03406468
Title: Re-Induction of a Systemic Immune Response After Initial Response With Immune Therapy With Radiotherapy in Metastatic or Locally Recurrent Lung Cancer
Brief Title: Re-Induction After Initial Response With Immune Therapy With Radiotherapy in Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: The Netherlands Cancer Institute (Other); Maastricht University Medical Center (Other); Zuyderland Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Re-Induction
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Non-Small Cell Carcinoma of Lung, TNM Stage 4
Keywords: non small cell lung cancer; immune therapy; radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Given the objective of this phase II trial and the limited number of patients, no formal statistical analyses are planned. Analysis will be limited to presentation of frequencies and proportions and the report of descriptive statistics (e.g. mean, median and/or range) in tabulated form.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy (Experimental): Patients continue the same immune therapy they already received and get radiotherapy to one lesion. The lesion may or may not be symptomatic. The preferred radiotherapy dose is 24 Gy in 3 fractions (dosage on the 10 Gy isodose is allowed), but other fractionation schedules (e.g. 30 Gy/ 10 fractions, 20 Gy/ 5 fractions, 20-24 Gy / 1 fraction for SRS (stereotactic radiosurgery)) are allowed if these are standard for a certain location or palliative indication in the body.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Patients continue the same immune therapy they already received and get radiotherapy to one lesion. The lesion may or may not be symptomatic. The preferred radiotherapy dose is 24 Gy in 3 fractions (dosage on the 10 Gy isodose is allowed), but other fractionation schedules (e.g. 30 Gy/ 10 fractions, 20 Gy/ 5 fractions, 20-24 Gy / 1 fraction for SRS (stereotactic radiosurgery)) are allowed if these are standard for a certain location or palliative indication in the body.

SUMMARY:
Radiotherapy in combination with different forms of immune therapy improved consistently local tumor control and very interestingly, lead to better systemic tumor control and the induction of specific anti-cancer immunity with a memory effect. In small series, it has been shown that a new long-lasting remission can be induced by irradiating one tumor site in patients who showed cancer progression after an initial response to immune therapy. In these series, the original immune therapy was continued and the treatment was very well tolerated. In this study the progression-free survival after radiotherapy to a single lesion will be investigated in patients with stage IV non-small cell lung cancer (NSCLC), who have at least achieved stable disease with immune therapy alone or concurrent immune therapy and chemotherapy.

DETAILED DESCRIPTION:
Radiation has consistently been shown to activate key elements of the immune system. Radiotherapy in combination with different forms of immune therapy such as anti-PD-(L)1, anti-CTLA4,immunocytokines, dendritic cell vaccination and Toll-like receptor agonists improved consistently local tumor control and very interestingly, lead to better systemic tumor control (the "abscopal" effect) and the induction of specific anti-cancer immunity with a memory effect. Moreover, as PD1/PD-L1 is upregulated by radiation and radiation can overcome resistance for PD-(L)1 blockage, their combination is logical.

In small series, it has been shown that a new long-lasting remission can be induced by irradiating one tumor site in patients who showed cancer progression after an initial response to immune therapy. In these series, the original immune therapy was continued and the treatment was very well tolerated. In this study the progression-free survival after radiotherapy to a single lesion will be investigated in patients with stage IV non-small cell lung cancer (NSCLC), who have at least achieved stable disease with immune therapy alone or concurrent immune therapy and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV non-small cell lung cancer
* Initially a Complete Remission, Partial Remission or Stable Disease under immune therapy alone or concurrent immune therapy and chemotherapy and now progressive disease
* Able to continue the immune therapy

Exclusion Criteria:

* Not able to continue the already initiated immune therapy
* Patients with any grade 3 toxocity
* Patients in whom radiotherapy cannot be delivered, according to the radiation oncologist at the multi-disciplinary patient discussion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 3 months after end of radiotherapy
  Progression free survival

SECONDARY OUTCOMES:
Remission rate irradiated lesion | 3 months after end of radiotherapy
  Remission rate (RECIST 1.0) of the irradiated lesion
Remission rate non-irradiated lesion(s) | 3 months after end of radiotherapy
  Remission rate (RECIST 1.0) of the non-irradiated lesion(s)
Toxicity | 3 months after end of radiotherapy
  Toxicity evaluation CTCAE4.0

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD, PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (3):
- Netherlands (3):
  - Zuyderland Hospital, Heerlen
  - Maastricht University Medical Center, Maastricht
  - MAATRO clinic, Maastricht

IPD SHARING:
Plan to Share IPD: No